CLINICAL TRIAL: NCT03648866
Title: A Thematic Analysis of the Effects of Compassion Rounds on Clinicians and the Families of NICU Patients
Brief Title: A Thematic Analysis of Compassion Rounds
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1320386
Record Dates: First submitted 2018-08-15; First posted 2018-08-28 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Spiritual Wellness
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Physicians: interview physicians who have conducted compassion rounds
  Interventions: Other: interview
- Chaplains: interview chaplains who have conducted compassion rounds
  Interventions: Other: interview
- Other Healthcare Providers: interview other healthcare providers who have conducted compassion rounds
  Interventions: Other: interview
- Patients: interview patients who have participated in compassion rounds
  Interventions: Other: interview
- Patient family members/friends: interview patient's loved ones who have participated with the patient in compassion rounds
  Interventions: Other: interview

INTERVENTIONS:
Other: interview — Initial interview and potential follow-up interviews and focus group with Florida Hospital employees.
  Interview participants in compassion rounds

SUMMARY:
The primary objective of this thematic analysis is to understand the experience of "Compassion Rounds" for patients, families, friends, and clinicians. The secondary objective of this study is to evaluate and interpret data to determine best practice recommendations for standardization and scalability.

DETAILED DESCRIPTION:
This research will be conducted as a Thematic Analysis. Participants will be recruited from those who take part in compassion rounds, including patients, their loved ones, physicians, chaplains, social workers, nurses, and other care providers.

Qualitative data on participants' experiences throughout the intervention will be collected and analyzed using thematic methodology. The data will be used to explain the psychosocial processes that influence participant experience and reported outcomes.

Qualitative methodology does not seek to verify hypotheses based on logical assumptions, as quantitative measures do, instead it is used to derive salient constructs directly from the data. This methodology allows inductive understanding of participants' social reality and perceptions of the treatment, resulting in explanations of how the treatment leads to outcomes and the identification of variables that may then be quantified for more generalizable study.

Semi-structured Interviews

Through semi-structured interviews, which will be recorded and transcribed, the researcher asks participants open-ended questions intended to elicit perspectives on their experience of compassion rounds, without limiting responses to pre-determined categories of interest. The following are examples:

"What/who do you remember most vividly?" "How would you describe your experience to a friend?" "What was most meaningful to you? "What made you feel uncomfortable?" "Would you do it again? Why or why not?" "What, if anything, changed after compassion rounding?"

Coding

The researcher codes and documents throughout data collection and analysis to lend transparency to the coding process and to keep a record of ideas to inform thematic exposition. The researcher assigns categorical codes (labels or concepts) to the transcribed responses line-by-line, analyzing patterns of relationships and using a constant comparison technique to identify similarities and differences throughout the data. The following coding techniques will be used to analyze transcriptions:

* open coding: the researcher segments the data into preliminary categories, based on similarity
* axial coding: the researcher groups the categories into themes that provide new ways of seeing and understanding the phenomenon under study
* selective coding: the researcher integrates the categories and themes to articulate a coherent theory of the phenomenon of study.

Theoretical Sampling Grounded theory research uses "theoretical sampling" to identify participants for interviews. Purposive samples are identified to initiate data collection and analysis, and to select participants who are likely to clarify, verify, or contradict data as it is collected. Sampling concludes when the data is "saturated," which occurs when coded categories are well-defined and no new significant insights are emerging from interviews.

Thematic Development and Validation

The researcher develops thematic explanations that stem from rendering participants' experiences throughout the practice of compassion rounding.

Themes are evaluated for fit and relevance and employee participants may be asked to validate the researcher's findings in follow-up interviews and focus groups.

Observation The researcher will also observe compassion rounding to collect data that will provide further insight to participants' experiences. Observations of interactions and reactions in real time will be documented and the data will be coded and analyzed using the techniques described above. Observational data will not be integrated into interview data, but will be used to confirm or contrast reported data.

ELIGIBILITY:
Inclusion Criteria:

1. An employee of Florida Hospital or Adventist Health System, or a physician with privileges there, or a patient, or a family or friend who has participated in compassion rounding at a Florida Hospital critical care unit
2. Over the age of 18
3. Able to provide informed consent
4. Must speak and understand English
5. Willing and able to provide a contact phone number

Exclusion Criteria:

1. Discernible cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from participants in compassion rounding, including patients, their loved ones, physicians, chaplains, social workers, nurses, and other care providers.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Validated Thematic Framework to Explain the Effects of Compassion Rounding | five months
  Analysis of data collected throughout the study will result in a validated theoretical framework to understand and explain the psychosocial processes that influence participant experience and reported outcomes.

SECONDARY OUTCOMES:
Compendium of Evidence-Based Best Practices for the Implementation of Compassion Rounding | five months
  Analysis of data collected throughout the study will result in an evidence-based compendium of best practices for the implementation of compassion rounding.

CONTACTS AND LOCATIONS:
Overall Officials: Kim McManus, Ph.D., Principal Investigator — FH Center for CREATION Health Research
Locations (1):
- AdventHealth Orlando, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No